CLINICAL TRIAL: NCT01468753
Title: Pilot Study: Acceptability, Feasibility and Efficacy of Vaginal Insemination in HIV Discordant Couples (Female Positive, Male Negative) Desiring Conception in Kisumu, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P30 AIO27763
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: HIV Discordant Couples
Keywords: Conception in HIV Discordant Couples; Reproduction in HIV Discordant Couples; Vaginal Insemination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Insemination (Experimental): Women will perform vaginal insemination during the fertile period of the menstrual cycle with the collected semen within one hour of collection. Vaginal insemination will occur within one hour of collection 2 days prior to ovulation, on the day of ovulation and 2 days after ovulation for up to 6 months or until conception occurs. For example, if ovulation were on day 14 of a 28 day menstrual cycle, vaginal insemination will occur on days 12, 14 and 16 of the cycle.
  Interventions: Procedure: Vaginal Insemination

INTERVENTIONS:
Procedure: Vaginal Insemination — Women will perform vaginal insemination during the fertile period with semen within one hour of collection. Vaginal insemination will occur within one hour of collection 2 days prior to ovulation, on the day of ovulation and 2 days after ovulation for up to 6 months or until conception occurs. For example, if ovulation were on day 14 of a 28 day menstrual cycle, vaginal insemination will occur on days 12, 14 and 16 of the cycle.

SUMMARY:
To evaluate the acceptability, feasibility, and efficacy of vaginal insemination as a method of conception in HIV discordant couples (female positive, male negative) desiring pregnancy in Kisumu, Kenya

DETAILED DESCRIPTION:
In sub-Saharan Africa, HIV is predominantly transmitted via discordant sexual relationships. With the availability of antiretroviral (ARV) medications, individuals infected with HIV can live relatively normal productive lives. Societal and cultural expectations as well as personal reproductive intentions drive HIV positive women in discordant relationships to conceive. Approximately 50% of HIV infected couples desire children. However, a safe and effective method of conception that minimizes the risk of sexual HIV transmission in HIV discordant couples with a positive woman and negative man has yet to be examined. To date, published studies have evaluated assisted reproductive methods in HIV discordant couples with a positive man to decrease the risk of HIV transmission. The investigators intend to evaluate the acceptability, feasibility and efficacy of vaginal insemination with semen for conception in HIV discordant (female positive, male negative) relationships in Kenya. In this pilot study, HIV discordant couples (female positive, male negative) desiring pregnancy will receive targeted reproductive counseling through the Safer and Healthy Conception Program for 6 months. This program will emphasize the consistent use of male condoms and teach couples assisted vaginal insemination for conception to minimize the risk of sexual HIV transmission.The investigators will compare the frequency of male condom use before and after intervention with an audio computer-assisted self-interview validated by random measurement of prostate specific antigen of vaginal secretions. The incidence of pregnancy following vaginal insemination will also be measured. The investigators hypothesize that our findings will provide evidence to support the routine use of vaginal insemination as a safe method of conception in HIV discordant couples (female positive, male negative). This pilot study is of significant public health importance because the use of vaginal insemination for conception in HIV discordant couples (female positive, male negative) is expected to reduce the likelihood of riskier sexual practices for childbearing and decrease the incidence of HIV in Sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* HIV discordant couple (female positive, male negative) desiring conception, monogamous relationship (minimum of three month duration), disclosure of HIV status to the sexual partner, women 18-34 years of age, sexually active (at least three encounters per month), expressed ability to consistently use male condoms, and follow the study protocol with respect to study visits and use of vaginal insemination.

Exclusion Criteria:

* pregnant (at the time of enrollment or run-in-period), women over 35 years of age (decreased fertility ≥ 35 years of age), self reported history of sterilization or infertility by either partner, use of teratogenic medication (e.g. Efavirenz), and clinical stage of HIV/AIDS 3 or 4.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of vaginal insemination in HIV discordant couples as compared to natural conception. | 8 months

SECONDARY OUTCOMES:
To evaluate the consistent use of male condoms for the prevention of sexual transmission of HIV. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Betty Njoroge, MB. ChB, MPH, Study Director — Kenya Medical Research Institute; Craig Cohen, MD, MPH, Study Chair — University of California, San Francisco
Locations (1):
- Family AIDS Care and Education Services - Lumumba Health Centre, Kisumu, Kenya